CLINICAL TRIAL: NCT07054944
Title: FEASIBILITY AND SAFETY OF INDOCYANINE GREEN (ICG) GUIDED SENTINEL LYMPH NODE MAPPING FOR PEDIATRIC SOLID TUMORS - T-LyM (Tumor-Lymph Node Mapping)
Brief Title: Tumor-Lymph Node Mapping
Acronym: T-LyM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Hafeez Abdel, Associate Professor - Department of Surgery, Pediatric Surgery (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00010277
Record Dates: First submitted 2025-06-18; First posted 2025-07-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Solid Tumors; Rhabdomyosarcoma; Sarcoma; Germ Cell Tumor
Keywords: PEDIATRIC CANCER
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma; Neoplasms, Germ Cell and Embryonal; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Indocyanine Green (ICG) and KARL STORZ ICG Imaging System (Experimental)
  Interventions: Diagnostic Test: ICG (Indocyanine Green)

INTERVENTIONS:
Diagnostic Test: ICG (Indocyanine Green) — Lymphatic mapping

SUMMARY:
The purpose of this study is to assess the feasibility and safety of ICG-guided intraoperative lymphography for detecting sentinel lymph nodes (SLN) in pediatric patients with solid tumors who require retroperitoneal lymph node dissection/sampling.

This trial is a single-site cross-sectional study. The injection of ICG directly into lymphatics draining the primary tumor will take place at the time of operation after the patient is under anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Any pediatric patient (under the age of 18 years) being treated at the University of Rochester Medical Center, Department of Surgery.
* Diagnosed with pediatric solid tumor
* Scheduled to undergo lymph node sampling as part of their clinical management.

Exclusion Criteria:

* Subjects with a history of iodide allergies.
* Inability or unwillingness of research participant or parent/legal guardian to give written informed consent.
* Currently pregnant.
* Infants under 650 grams.
* Patients with extensive prior surgery at the primary site or nodal basin expected to affect the lymphatic drainage.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients with Successful Sentinel Lymph Node (SLN) Detection Using ICG Fluorescence | Baseline
  Success is defined as the intraoperative identification of at least one fluorescent sentinel lymph node (SLN) after indocyanine green (ICG) injection using an Iridium system optimized for near-infrared detection. Visualization of the SLN indicates uptake of ICG within the lymphatic basin.

OTHER OUTCOMES:
Accuracy of SLN Biopsy as Measured by Concordance Between SLN Pathology and Nodal Basin Pathology | During surgery (Day 0), based on intraoperative and postoperative pathology reports finalized within 7 days
  Accuracy is assessed by comparing the pathology results of the SLN and the retroperitoneal lymph node basin dissection. True positives and true negatives are defined as SLN and nodal basin showing matching tumor status (both positive or both negative). Discordant finding is defined as tumor basin positive for tumor while SLN is negative for tumor. Discordant findings are considered false negatives. A tumor positive SLN in a tumor negative nodal basin is not considered discordant or false positive because sentinel may be the first and only tumor involved lymph node within the nodal basin.